CLINICAL TRIAL: NCT02540148
Title: Transpalpebral Micro-Current Electrical Stimulation for the Treatment of Dry Age-Related Macular Degeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Eye Machine Canada Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NO001D
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Age-Related (Dry) Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Active Treatment (Experimental): Patients will be fully consented before the start of the study. In the treatment group, subjects will undergo a treatment session to the enrolled eyes for three days during Week 1, followed by a single treatment session during Weeks 2, 14 and 26 with the Nova Oculus device. A treatment session is 15 minutes of treatment on each closed eye lid for a total of 30 minutes. ETDRS visual acuity will be performed on all subjects at enrollment (prior to the first treatment), prior to each treatment session, and at four weeks from enrollment. The effect of treatments with the Nova Oculus device compared to sham treatment on the visual acuity of subjects with dry AMD will be determined.e.
  Interventions: Device: Nova Oculus™ Micro-current electrical stimulation
- Non-active treatment (Sham Comparator): A second group of subjects will act as the control group. This group will undergo sham treatment to the enrolled eyes at the same intervals as the treatment group (Weeks 2, 14 and 26), but with a nonfunctional Nova Oculus device. A treatment session is 15 minutes of treatment on each closed eye lid for a total of 30 minutes. ETDRS visual acuity will be performed on all subjects at enrollment (prior to the first treatment), prior to each treatment session, and at four weeks from enrollment. The effect of treatments with the Nova Oculus device compared to sham treatment on the visual acuity of subjects with dry AMD will be determined.
  Interventions: Device: Nova Oculus™ Micro-current electrical stimulation - Sham treatment

INTERVENTIONS:
Device: Nova Oculus™ Micro-current electrical stimulation — Active treatment with transpalpebral micro-current electrical stimulation device, 3 sessions within 5 days of the 1st treatment. 1 session during weeks 2, 14 and 26.
  Arms: Active Treatment
Device: Nova Oculus™ Micro-current electrical stimulation - Sham treatment — Non-active treatment with transpalpebral micro-current electrical stimulation SHAM device, 3 sessions within 5 days of the 1st treatment. 1 session during weeks 2, 14 and 26.
  Arms: Non-active treatment

SUMMARY:
Assess the effectiveness of externally applied micro current electrical stimulation on improving the ETDRS visual acuity in subjects with vision loss from dry age-related macular degeneration (AMD)

DETAILED DESCRIPTION:
Micro-current electrical stimulation will be used to treat /each eye in a group of subjects with dry AMD. 60 subjects will be randomly divided into two groups. A ratio of 1:3 will be maintained between control and the experimental groups. In the treatment group, subjects will undergo a treatment session to the enrolled eyes daily for three days during week 1, followed by a single treatment session during weeks 2, 14 and 26 with the Nova Oculus device. A second group of subjects will act as the control group. This group will undergo sham treatment at the same treatment intervals with a non-functional Nova Oculus device. ETDRS visual acuity will be performed on all subjects at enrollment prior to each treatment and at four weeks from enrollment. The effect of treatments with the Nova Oculus device compared to sham treatment on the ETDRS visual acuity of subjects with dry AMD will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Fifty years of age or older
* Male or female
* Best-corrected vision 20/50 to 20/200 for each enrolled eye
* Confirmed diagnosis of dry AMD
* Vision loss attributable to dry AMD
* Subjects must be highly motivated, alert, oriented, mentally competent and able to understand and comply with the requirements of the study, abide by the restrictions, return for all required visits, and provide voluntary informed consent

Exclusion Criteria:

* Any visually significant retinal pathology other than dry AMD
* Previous intravitreal injection
* Seizure disorders
* Previous vitreo-retinal surgery. (ERM, PPV, RD etc)
* Dense cataract
* Eyelid pathology at the treatment sites
* Glaucoma patients with a visual field mean defect of greater than 10dB on Humphrey visual field testing
* Glasses are up to date (prescription <1 year old)
* Any prior electrical micro-stimulation treatment to the eyes
* Poor general health
* Active cancer
* Life expectancy less than 12 months
* Non-ambulatory
* Not considered suitable for participation for any other reason

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Measure the increase in ETDRS visual acuity for those treated with Nova Oculus™ device to control subjects who did not receive active treatment. | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Parkinson, MD, Principal Investigator — Independent
Locations (1):
- Dr. Kevin Parkinson, Coquitlam, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parkinson KM, Sayre EC, Tobe SW. Evaluation of visual acuity in dry AMD patients after microcurrent electrical stimulation. Int J Retina Vitreous. 2023 Jun 18;9(1):36. doi: 10.1186/s40942-023-00471-y. PMID 37331928